CLINICAL TRIAL: NCT06802614
Title: A Randomized Controlled Clinical Trial Comparing the Efficacy of Two Experimental Bleaching Gels With and Without Nanoparticles and Light Irradiation Versus Whiteness HP 35% and Whiteness HP AutoMixx 6% in Patients With A2-C4 Tooth Discolorations
Brief Title: Efficacy and Safety Assessment of Experimental Bleaching Agents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OUCOD001
Record Dates: First submitted 2025-01-17; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Tooth Discoloration; Dentin Sensitivity; Patient Satisfaction
Keywords: Tooth Whitenining; Dental Bleaching; Hydrogen Peroxide; Titanium Dioxide Nanoparticles
MeSH Terms: conditions — Tooth Discoloration; Dentin Sensitivity; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: This will be a randomized, parallel-arm clinical trial that compares the efficacy of the two experimental bleaching gels, with and without nanoparticles, versus two commercial products that serve as the control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- 1. Gel A with nanoparticles, no light. (Experimental): An experimental Bleaching Gel composed of Carbomer 940 hydrogel + 6% Hydrogen Peroxide + 5% nanoparticles (NF_TiO₂) will be applied for 50 minutes.
  Interventions: Device: BLEACHING GEL A; Device: 5% NF_TiO2
- 2. Gel A with nanoparticles, with light. (Experimental): An experimental Bleaching Gel composed of Carbomer 940 hydrogel + 6% Hydrogen Peroxide + 5% nanoparticles (NF_TiO₂) + 405 nm violet LED light will be applied for 50 minutes after the gel is applied.
  Interventions: Device: BLEACHING GEL A; Device: 5% NF_TiO2; Radiation: VISIBLE LIGHT IRRADIATION
- 3. Gel A without nanoparticles, no light. (Experimental): An experimental Bleaching Gel composed of Carbomer 940 hydrogel + 6% Hydrogen Peroxide will be applied for 50 minutes.
  Interventions: Device: BLEACHING GEL A
- 4. Gel A without nanoparticles, with light. (Experimental): An experimental Bleaching Gel composed of Carbomer 940 hydrogel + 6% Hydrogen Peroxide + 405 nm violet LED light applied for 50 minutes.
  Interventions: Device: BLEACHING GEL A; Radiation: VISIBLE LIGHT IRRADIATION
- 5. Gel B with nanoparticles, no light. (Experimental): Hyaluronic Acid hydrogel + 6% Hydrogen Peroxide + 5% nanoparticles (NF_TiO₂) applied for 50 minutes.
  Interventions: Device: 5% NF_TiO2; Device: BLEACHING GEL B
- 6. Gel B with nanoparticles, with light. (Experimental): Hyaluronic Acid hydrogel + 6% Hydrogen Peroxide + 5% nanoparticles (NF_TiO₂) + 405 nm violet LED light applied for 50 minutes.
  Interventions: Device: 5% NF_TiO2; Device: BLEACHING GEL B; Radiation: VISIBLE LIGHT IRRADIATION
- 7. Gel B without nanoparticles, no light. (Experimental): Hyaluronic Acid hydrogel + 6% Hydrogen Peroxide applied for 50 minutes.
  Interventions: Device: BLEACHING GEL B
- 8. Gel B without nanoparticles, with light. (Experimental): Hyaluronic Acid hydrogel + 6% Hydrogen Peroxide + 405 nm violet LED light applied for 50 minutes.
  Interventions: Device: BLEACHING GEL B; Radiation: VISIBLE LIGHT IRRADIATION
- 9. Whiteness HP 35% no light (control). (Active Comparator): Whiteness HP 35% applied for 30 minutes.
  Interventions: Device: Whiteness HP 35%
- 10. Whiteness HP 35% with light (control). (Active Comparator): Whiteness HP 35% + 405 nm violet LED light applied for 30 minutes.
  Interventions: Radiation: VISIBLE LIGHT IRRADIATION; Device: Whiteness HP 35%
- 11. Whiteness HP AutoMixx 6% no light (control) (Active Comparator): Whiteness HP AutoMixx 6% applied for 30 minutes.
  Interventions: Device: Whiteness HP Automixx 6%
- 12. Whiteness HP AutoMixx 6% with light (control) (Active Comparator): Whiteness HP 6% + 405 nm violet LED light applied for 30 minutes.
  Interventions: Radiation: VISIBLE LIGHT IRRADIATION; Device: Whiteness HP Automixx 6%

INTERVENTIONS:
Device: BLEACHING GEL A — Carbomer 940 hydrogel + 6% Hydrogen Peroxide
  Arms: 1. Gel A with nanoparticles, no light.; 2. Gel A with nanoparticles, with light.; 3. Gel A without nanoparticles, no light.; 4. Gel A without nanoparticles, with light.
Device: 5% NF_TiO2 — Bioactive nanoparticles
  Arms: 1. Gel A with nanoparticles, no light.; 2. Gel A with nanoparticles, with light.; 5. Gel B with nanoparticles, no light.; 6. Gel B with nanoparticles, with light.
Device: BLEACHING GEL B — Hyaluronic Acid hydrogel + 6% Hydrogen Peroxide
  Arms: 5. Gel B with nanoparticles, no light.; 6. Gel B with nanoparticles, with light.; 7. Gel B without nanoparticles, no light.; 8. Gel B without nanoparticles, with light.
Radiation: VISIBLE LIGHT IRRADIATION — Low intensity visible light irradiation (405 nm)
  Arms: 10. Whiteness HP 35% with light (control).; 12. Whiteness HP AutoMixx 6% with light (control); 2. Gel A with nanoparticles, with light.; 4. Gel A without nanoparticles, with light.; 6. Gel B with nanoparticles, with light.; 8. Gel B without nanoparticles, with light.
Device: Whiteness HP 35% — Commercially available bleaching gel
  Arms: 10. Whiteness HP 35% with light (control).; 9. Whiteness HP 35% no light (control).
Device: Whiteness HP Automixx 6% — Commercially available bleaching gel
  Arms: 11. Whiteness HP AutoMixx 6% no light (control); 12. Whiteness HP AutoMixx 6% with light (control)

SUMMARY:
Tooth bleaching is widely used to treat the colors of teeth. This study compares the efficiency of two experimental bleaching gels, with and without nanoparticles, and with and without light activation versus two commercial bleaching products of low and high concentrations. The objective is to evaluate tooth color change, sensitivity, and patient satisfaction in patients with moderate yellowing of their teeth. Methods: This is a randomized controlled trial that will include 120 participants aged 18-65 years. Participants will be randomly assigned to one of 12 treatment groups: Gel A (with or without nanoparticles, with or without light), Gel B (with or without nanoparticles, with or without light), Whiteness HP 35% (with or without light) and Whiteness Automixx 6% (with or without light). The primary outcome is tooth color change, measured using a commercially-available equipment. Secondary outcomes will include tooth sensitivity and patient satisfaction. Randomization will be computer-generated. Results: The study is expected to show differences in color change between the experimental and commercial gels. Tooth sensitivity and patient satisfaction will be evaluated to determine the overall effectiveness and safety of the treatments. Conclusions: This trial will provide information into the whitening efficacy of two experimental gels compared to two widely used commercial products.

DETAILED DESCRIPTION:
Tooth whitening treatments are widely used to address dental discoloration. This study compares the efficacy of two experimental bleaching gels, Gel A (Carbomer 940 + 6% Hydrogen Peroxide) and Gel B (Hyaluronic Acid + 6% Hydrogen Peroxide), with and without 5% of NF_TiO₂ nanoparticles, and with and without light activation (405 nm, 30 min) versus a control bleaching product (Whiteness HP 35%, FGM). The aim is to evaluate tooth color change, sensitivity, and patient satisfaction in patients with baseline tooth discoloration ranging from shades A3 to C4 on the Vita Classical Shade Guide. Methods: This is a randomized controlled trial that will include 200 participants aged 18-65 years with mild to moderate tooth discoloration. Participants will be randomly assigned to one of 10 treatment groups: Gel A (with or without nanoparticles, with or without light), Gel B (with or without nanoparticles, with or without light), Whiteness HP 35% (with or without light) and Whiteness Automixx 6% (with or without light). The primary outcome is tooth color change, measured using the Vita EasyShade V system to assess ΔE, ΔE00, and Whiteness Index for Dentistry (WiD). Secondary outcomes will include tooth sensitivity (measured with a Visual Analog Scale) and patient satisfaction (assessed via post-treatment questionnaire). Randomization will be computer-generated, and the study will be double-blinded for evaluators. Results: The study is expected to detect significant differences in color change between the experimental gels and Whiteness HP 35%, with or without nanoparticles and light activation. Tooth sensitivity and patient satisfaction will be evaluated to determine the overall effectiveness and safety of the treatments. Conclusions: This trial will provide insights into the whitening efficacy of two experimental gels compared to a widely used commercial product. The inclusion of nanoparticles and light activation as variables will help determine the optimal conditions for effective tooth bleaching in patients with moderate discoloration. The results will contribute to evidence-based recommendations for aesthetic dental treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years old.
* Healthy periodontal tissues.
* Willingness to participate and follow the post-treatment protocols.
* Ability to provide informed consent.
* Teeth having baseline colors ranging from shade A2 to C4

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Teeth with restorations.
* History of dentin hypersensitivity.
* Active caries, periodontal disease or endodontically treated teeth.
* Use of substances that could affect tooth color during the trial, such as smoking and vaping.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Tooth Color - Delta E | At baseline (T0), after each clinical session (T1, T2 and T3; 7 days interval between sessions) and at T4 (14 days after T3)
  Delta E ; This outcome measure is dimensionless and will be extracted from L*, a* and b* values.
Tooth Color - Delta E00 | At baseline (T0), after each clinical session (T1, T2 and T3; 7 days interval between sessions) and at T4 (14 days after T3)
  Delta E00; This outcome measure is dimensionless and will be extracted from L*, a* and b* values.
Tooth Color - WiD | At baseline (T0), after each clinical session (T1, T2 and T3; 7 days interval between sessions) and at T4 (14 days after T3)
  WiD; This outcome measure is dimensionless and will be extracted from L*, a* and b* values.

SECONDARY OUTCOMES:
Tooth sensitivity | At baseline (T0), after each clinical session (T1, T2 and T3; 7 days interval between sessions) and at T4 (14 days after T3)
  Visual Analog Scale (VAS). The scale will vary from 0 (no pain) to 10 (worst pain possible). In this outcome measure, higher scores reflect outcomes that are worse in nature
Patient Satisfaction | at T4 (14 days after T3)
  Post-treatment questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando L Esteban Florez, D.D.S., M.S., Ph.D., Principal Investigator — The University of Oklahoma Health Sciences Center College of Dentistry
Locations (1):
- The University of Oklahoma Health Sciences Center College of Dentistry, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
We will not share individual data. We plan on sharing data that have been statistically analyzed. The sharing of this data will occur via peer-reviewed publications and conferences such as the annual meetings of the American Association for Dental, Oral and Craniofacial Research, the International Association for Dental Research and the annual meeting of the Academy of Dental Materials.

REFERENCES:
- [Background] Kury M, Hiers RD, Zhao YD, Picolo MZD, Hsieh J, Khajotia SS, Esteban Florez FL, Cavalli V. Novel Experimental In-Office Bleaching Gels Containing Co-Doped Titanium Dioxide Nanoparticles. Nanomaterials (Basel). 2022 Aug 30;12(17):2995. doi: 10.3390/nano12172995. PMID 36080033
- [Background] Matos ICRT, Kury M, de Melo PBG, de Souza LVS, Esteban Florez FL, Cavalli V. Effects of experimental bleaching gels containing co-doped titanium dioxide and niobium pentoxide combined with violet light. Clin Oral Investig. 2023 Aug;27(8):4827-4841. doi: 10.1007/s00784-023-05113-z. Epub 2023 Jun 28. PMID 37369816
- [Background] Kury M, Esteban Florez FL, Tabchoury CPM, Cavalli V. Effects of experimental in-office bleaching gels incorporated with co-doped titanium dioxide nanoparticles on dental enamel physical properties. Odontology. 2025 Jan;113(1):318-330. doi: 10.1007/s10266-024-00976-4. Epub 2024 Jul 4. PMID 38963521
- [Background] Kury M, de Oliveira Ribeiro RA, de Souza Costa CA, Florez FLE, Cavalli V. Co-doped titanium dioxide nanoparticles decrease the cytotoxicity of experimental hydrogen peroxide gels for in-office tooth bleaching. Clin Oral Investig. 2024 Sep 25;28(10):550. doi: 10.1007/s00784-024-05916-8. PMID 39320486